CLINICAL TRIAL: NCT01192841
Title: Physician Dress Code And Microbial Colonization Of The White Coat: Does Physician Dress Code Alter Bacterial Colonization Rate On The Clothing Of Physicians?
Brief Title: Bacterial Contamination of Workwear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Marisha Burden, MD, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-1137
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Bacterial Contamination of Physician Attire
Keywords: physician uniform; MRSA; bacterial contamination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- White coat group (No Intervention): Participants continued their regular practice of wearing their physician white coat.
- Uniform group (Experimental): Participants were given a clean uniform (scrubs) at the beginning of the day.
  Interventions: Other: Physician uniform

INTERVENTIONS:
Other: Physician uniform — Participants were given a clean uniform (scrubs) on the day of the study. They wore this for approximately 8 hours.
  Arms: Uniform group

SUMMARY:
Governmental agencies in the United Kingdom and Scotland have recently instituted guidelines banning physicians' white coats and wearing of long-sleeved garments to decrease hospital transmission of bacteria. The purpose of this study is to compare the bacterial contamination of physicians' white coats with that of newly laundered, standardized short-sleeved uniforms after an eight-hour workday and to determine the rate at which bacterial contamination of the uniform ensues. Our hypothesis was that the physician white coat would have more bacterial contamination at the end of the work day.

DETAILED DESCRIPTION:
Governmental agencies in the United Kingdom and Scotland have recently instituted guidelines banning physicians' white coats and wearing of long-sleeved garments to decrease nosocomial transmission of bacteria. Our goal was to compare the degree of bacterial and methicillin-resistant Staphylococcus aureus contamination of physicians' white coats with that of newly laundered, standardized short-sleeved uniforms after an eight-hour workday and to determine the rate at which bacterial contamination of the uniform ensues. 100 interns, residents, and hospitalists on an internal medicine service were randomized to wear either physician white coat or newly laundered, short-sleeved uniform. Bacterial colony counts and the frequency with which methicillin-resistant Staphylococcus aureus was found was compared in the two groups and over time. Our initial hypothesis was that physician white coats would have more bacterial contamination at the end of the work day.

ELIGIBILITY:
Inclusion Criteria:

* Internal medicine interns, residents, and hospitalists working on acute medicine ward service.

Exclusion Criteria:

* Not willing/unable to participate in study
* Not working a full 8 hour day in the hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Bacterial colony counts and the frequency with which methicillin-resistant Staphylococcus aureus was found over time | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marisha Burden, MD, Principal Investigator — Denver Health and Housing Authority
Locations (1):
- Denver Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Burden M, Cervantes L, Weed D, Keniston A, Price CS, Albert RK. Newly cleaned physician uniforms and infrequently washed white coats have similar rates of bacterial contamination after an 8-hour workday: a randomized controlled trial. J Hosp Med. 2011 Apr;6(4):177-82. doi: 10.1002/jhm.864. Epub 2011 Feb 10. PMID 21312328